CLINICAL TRIAL: NCT00902083
Title: Open-Label, Multi-Center, Randomized, Active-Controlled, Phase 4 Study of rAd-p53 Gene Mono-Therapy, With Concurrent Chemotherapy, or Combination With Surgery in Subjects With Advanced Oral and Maxillofacial Malignant Tumors
Brief Title: rAd-p53 Gene Therapy for Advanced Oral and Maxillofacial Malignant Tumors
Acronym: rAd-p53
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shenzhen SiBiono GeneTech Co.,Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: rAd-p53-002
Record Dates: First submitted 2009-05-11; First posted 2009-05-14 (Estimated); Last update posted 2012-04-09 (Estimated); Status verified 2010-02

CONDITIONS: Advanced Oral and Maxillofacial Malignant Tumors
Keywords: p53 gene; Oral and Maxillofacial; gene therapy; malignant tumors
MeSH Terms: conditions — Neoplasms | interventions — Genes, p53; Surgical Procedures, Operative; Drug Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- surgery plus p53 gene (Experimental): using p53 gene therapy before surgery
  Interventions: Drug: p53 gene with surgery
- surgery alone (Active Comparator): Surgery without pre-p53 gene therapy
  Interventions: Procedure: surgery
- p53 plus chemotherapy (Experimental): p53 gene therapy with concurrent chemotherapy
  Interventions: Drug: p53 with chemotherapy
- p53 gene therapy alone (Experimental): Intra-tumor injectio of rAd-p53 gene with no concurrent treatment
  Interventions: Drug: p53 gene therapy

INTERVENTIONS:
Drug: p53 gene with surgery — pre-surgery p53 gene treatment: 10exp12 virus particles per 3 days for 5 times
  Other Names: no other names
  Arms: surgery plus p53 gene
Procedure: surgery — remove tumor surgery
  Other Names: no other names
  Arms: surgery alone
Drug: p53 with chemotherapy — p53 gene treatment: 10exp12 virus particles per 3 days for 10 times Chemotherapy: standard chemotherapy
  Other Names: no other names
  Arms: p53 plus chemotherapy
Drug: p53 gene therapy — p53 gene treatment: 10exp12 virus particles per 3 days for 10 times
  Other Names: no other names
  Arms: p53 gene therapy alone

SUMMARY:
This is multicenter, open-label, randomized, active-controled, phase IV study of local direct intra-tumor injection of rAd-p53 monotherapy, with concurrent chemotherapy , or combination with surgery for treatment of advanced oral and maxillofacial malignant tumors.

DETAILED DESCRIPTION:
Primary objectives of this study is to determine the efficacy profiles of rAd-p53 intra-tumor injection alone, with concurrent chemotherapy, or combination with surgery for treatment of advanced oral and maxillofacial malignant tumors(stage III or IV) including target lesion complete response rate (LCR) and overall target lesion response rate (OLR), response duration (RD), and progress-free survival (PFS).

The secondary objectives of this study is to investigate overall response rate (OPCR) and overall complete response rate (OCR), overall survival (OS), ECOG, and safety of rAd-p53 monotherapy and combined with chemotherapy,or surgery.

ELIGIBILITY:
Inclusion Criteria:

1. Advanced stages of Oral and Maxillofacial malignant tumors (stage III and VI)
2. At least one target tumor can be injected with study drug, the largest diameter greater than 2 cm
3. Histologically confirmed Oral and Maxillofacial malignant tumors
4. No prior chemotherapy, radiotherapy or biological tumor therapy in 2 weeks
5. Age: 18-85 years old
6. Expected to survive more 12 weeks
7. ECOG:0-2
8. Neutrophils≥1.5×109/L,Platelet≥ 80×109/L, Hb≥80g/L, bilitubin≤2mg/dl,ALT and AST ≤2×institutional upper limit of normal, Cr ≤1.5×institutional upper limit of normal,coagulation tests (PTT and INR) within normal range
9. Subject provided signed informed consent

Exclusion Criteria:

1. Hypersensitive to study drug
2. Tumor(s) locate very close to important blood vessels and nerves, which affect injection
3. With a coagulation and bleeding disorder
4. With uncontrolled, intercurrent illness including but limited to symptomatic neurological illness, symptomatic congestive heart failure, unstable angina pectoris, significant pulmonary disease or hypoxia, or psychiatric illness
5. Local infection close to injection site or systemic infection
6. Pregnant or lactating
7. Principle investigator consider not suitable -

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 600 (Estimated)
Dates: Start 2009-06; Primary Completion 2012-07 (Estimated); Study Completion 2012-07 (Estimated)

PRIMARY OUTCOMES:
overall best response rate | 3 years

SECONDARY OUTCOMES:
progress free survival | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Longjiang Li, PhD, MD, Principal Investigator — West China Hospital
Locations (1):
- West China Hospital, Sichuan University, Chengdu, Sichuan, China